CLINICAL TRIAL: NCT05515445
Title: Study to Evaluate the Pharmacokinetics of Chiglitazar in Subjects With Hepatic Impairment and Normal Hepatic Function
Brief Title: Pharmacokinetics of Chiglitazar in Subjects With Hepatic Impairment and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGZ108
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — chiglitazar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Experimental): Subjects with normal hepatic function will receive a single 48 mg oral dose of Chiglitazar
  Interventions: Drug: Chiglitazar
- Mild Hepatic Impairment (Experimental): Subjects with mild hepatic impairment will receive a single 48 mg oral dose of Chiglitazar
  Interventions: Drug: Chiglitazar
- Moderate Hepatic Impairment (Experimental): Subjects with moderate hepatic impairment will receive a single 48 mg oral dose of Chiglitazar
  Interventions: Drug: Chiglitazar
- Severe Hepatic Impairment (Experimental): Subjects with severe hepatic impairment will receive a single 48 mg oral dose of Chiglitazar
  Interventions: Drug: Chiglitazar

INTERVENTIONS:
Drug: Chiglitazar — Oral single dose 48 mg

SUMMARY:
This Phase 1 open label study is being conducted to directly characterize the pharmacokinetic (PK) profiles of Chiglitazar following administration of a single oral dose in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent, able to comply with the requirements of the study.
* Male or female, between 18 and 79 years of age.
* 18≤BMI≤30. Weight of male ≥50 kg and Weight of female ≥ 45 kg.
* No medication within 2 weeks, or stable medication for at least 4 weeks prior to screening.
* Physical examination, vital signs examination, 12-lead electrocardiogram (ECG) examination, and laboratory test have been determined by the investigator to be suitable for participating in this trial.

Exclusion Criteria:

* Allergic constitution, or allergic to PPAR agonist drugs or any component of Chiglitazar tablets.
* received PPAR agonist drugs within 2 weeks before screening.
* Those who have been vaccinated within 4 weeks before screening, or who plan to be vaccinated during the trial.
* positive test for COVID-19, TP antibody and RPR, or HIV antibody.
* suffer from uncontrolled serious diseases of cardiovascular, respiratory, gastrointestinal, endocrine, blood, mental/nervous systems within 1 year before screening.
* have previously undergone surgery that may affect the absorption, distribution, metabolism, and excretion of drugs; anticipate surgery or hospitalization during the trial.
* Drug abusers, or positive test for drugs of abuse.
* Smoking more than 5 cigarettes per day on average within 3 months before screening.
* The average daily alcohol intake in the 3 months prior to screening exceeds the following criteria: more than 14 g for women, or more than 28 g for men; ingested any products containing alcohol within 48 hours before administration; positive alcohol breath test; patients with alcoholic cirrhosis who did not abstinence within 3 months before screening.
* Ingestion of grapefruit juice/grapefruit juice, food or drink rich in methylxanthine within 48 hours before administration; strenuous exercise or other factors that affect drug absorption, distribution, metabolism, excretion.
* participated in clinical trials of any drug or medical device within 3 months before screening.
* donated blood (or blood loss) ≥400 mL within 3 months before screening, or received whole blood or red blood cell suspension.
* Female subjects who are breastfeeding or positive test of serum pregnancy.
* eGFR<60 mL/min/1.73m2.
* Other circumstances assessed by the investigator are not suitable for participating in this trial.

Supplementary exclusion criteria for subjects with hepatic impairment：

* drug-induced liver injury.
* acute liver function damage caused by various reasons;
* complications of liver cirrhosis that the investigator considers inappropriate to participate in the study.
* diseases that seriously affect bile excretion.

Supplementary exclusion criteria for subjects with normal hepatic function:

* history of hepatic function damage, or who may have hepatic function damage that the investigator considers to be clinically significant.
* positive test for HBsAg, HCV.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Cmax | 4 days
  Maximum plasma concentration
AUC0-t and AUC0-inf | 4 days
  Area under of the curve (AUC0-t and AUC0-inf)

CONTACTS AND LOCATIONS:
Overall Officials: LiYan Miao, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China